CLINICAL TRIAL: NCT07317726
Title: Recent Trends in Stage Migration of Gastrointestnial Carcinoid Tumors Over Two Decades: a Retrospective SEER-based Analysis 2000-2022
Status: Completed | Type: Observational
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, asmaa salama ibrahim, Resident physician of gastroenterology, Suez Canal University
Other Study IDs: A278
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Carcinoid Tumor; SEER Database Analysis; Stage
MeSH Terms: conditions — Carcinoid Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Stage migration occurs when patients sound to have better survival or increased incidence rates at the early stage at diagnosis due to early detection of the disease. As carcinoid tumors are rare and there are no data supporting stage migration, the aim of this study was to perform comprehensive trends analysis in addition to survival analysis over two decades.

ELIGIBILITY:
Inclusion Criteria:

* patients with gastrointestinal carcinoid tumors

Exclusion Criteria:

* patients with unknown age data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: the investigators analyzed the data from cancer registries participating in Surveillance, Epidemiology, and End Results (SEER) software for patients diagnosed with primary GI carcinoid tumors from 2000-2022 using a rate session to calculate the percent change and annual percent change in addition to incidence rates.
Sampling Method: Probability Sample
Enrollment: 93481 (Actual)
Dates: Start 2000-12-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
The percent change and annual percent change for gastrointestinal carcinoids | 2000-2022
the percent change and annual percent change for gastrointestinal carcinoids across different stage distribution at diagnosis (localized, regional, distant, unknown) | 2000-2022

IPD SHARING:
Plan to Share IPD: Undecided